CLINICAL TRIAL: NCT03291171
Title: A Randomized Controlled Trial to Identify the Effect and the Working Mechanisms of MyPlan 2.0, a Self-regulation-based e- and mHealth Intervention Targeting Physical Activity and Sedentary Behaviour, in Adults With Type 2 Diabetes.
Brief Title: Identifying the Effect and Working Mechanisms of MyPlan 2.0 in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyPlan2.0_diabetes
Record Dates: First submitted 2017-09-11; First posted 2017-09-25 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Chronic Disease
Keywords: physical activity; sedentary behaviour; type 2 diabetes; eHealth; mHealth; self-regulation; behaviour change techniques
MeSH Terms: conditions — Chronic Disease; Motor Activity; Diabetes Mellitus, Type 2; Self-Control

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: intervention group and waiting-list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the e- and mHealth intervention 'MyPlan 2.0'.
  Interventions: Behavioral: MyPlan 2.0
- Waiting-list control group (No Intervention): Participants will not receive the e- and mHealth intervention 'MyPlan 2.0', but will be given access to the intervention after all testing phases.

INTERVENTIONS:
Behavioral: MyPlan 2.0 — MyPlan 2.0 consists of five sessions. During these five sessions the following behaviour change techniques are used to motivate users to be more physically active or to sit less: exploring risk perceptions and perceived benefits, exploring social support, providing feedback, action planning, coping planning and monitoring.
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate whether and how 'MyPlan 2.0' helps adults with type 2 diabetes to be more physically active or less sedentary. Two groups will be created, an intervention group and a waiting-list control group.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether and how 'MyPlan 2.0' helps adults with type 2 diabetes to be more physically active or less sedentary. Two groups will be created, an intervention group and a waiting-list control group. Both groups will be tested during three testing waves: pretest, posttest and follow-up test. Only the intervention group will be given acces to 'MyPlan 2.0'. 'MyPlan 2.0' consists of a website and mobile application targeting physical activity and sedentary behaviour. The intervention has a duration of five weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Type 2 diabetes
* Have access to internet
* Being computer literate

Exclusion Criteria:

* not Dutch Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in objective total, light and moderate-to-vigorous physical activity (PA) | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total, light and moderate-to-vigorous physical activity, measured via accelerometers
Change in objective sedentary behaviour | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total sitting time, measured via accelerometers
Change in self-reported total, light and moderate-to-vigorous physical activity (PA) | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total, light and moderate-to-vigorous physical activity, measured via the International Physical Activity Questionnaire (IPAQ)
Change in self-reported sedentary behaviour | Pretest, posttest (6 weeks) and follow-up (6 months)
  Change in amount of total sitting time, measured via the LASA sedentary behaviour self-report questionnaire

SECONDARY OUTCOMES:
Change in self-efficacy | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Change in amount of self-efficacy to change behaviour, measured via 3 validated items (questionnaire)
Change in outcome expectancies | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Outcome expectancies regarding the behaviour change, measured via 3 validated items (questionnaire)
Change in risk perception | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Risk perception about the behaviour, measured via 3 validated items (questionnaire)
Change in intention | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Amount of intention to change the behaviour, measured via 3 validated items (questionnaire)
change in action planning | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Amount of action planning for behaviour change, measured via 3 validated items (questionnaire)
change in coping planning | Pretest, after week 1, after week 2, after week 3, after week 4, posttest (6 weeks), and follow-up (6 months)
  Amount of coping planning for behaviour change, measured via 3 validated items (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Ilse De Bourdeaudhuij, Professor, Principal Investigator — University Ghent; Geert Crombez, Professor, Principal Investigator — University Ghent; Maïté Verloigne, PostDoc, Principal Investigator — University Ghent
Locations (1):
- Department of Movement and Sports Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poppe L, De Bourdeaudhuij I, Verloigne M, Shadid S, Van Cauwenberg J, Compernolle S, Crombez G. Efficacy of a Self-Regulation-Based Electronic and Mobile Health Intervention Targeting an Active Lifestyle in Adults Having Type 2 Diabetes and in Adults Aged 50 Years or Older: Two Randomized Controlled Trials. J Med Internet Res. 2019 Aug 2;21(8):e13363. doi: 10.2196/13363. PMID 31376274